CLINICAL TRIAL: NCT03895970
Title: Lenvatinib Combined Pembrolizumab as a Second-line Treatment in Advanced Hepatobiliary Tumors: a Single-center, Single-arm, Non-randomized Clinical Study
Brief Title: Lenvatinib Combined Pembrolizumab in Advanced Hepatobiliary Tumors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JS-1864
Record Dates: First submitted 2019-03-28; First posted 2019-03-29 (Actual); Last update posted 2023-03-29 (Actual); Status verified 2022-11

CONDITIONS: Liver Neoplasm Malignant Primary; Cholangiocarcinoma; Combinational Immunotherapy; Biomarker
Keywords: Hepatobiliary Cancer; Pembrolizumab; Lenvatinib; Biomarker
MeSH Terms: conditions — Cholangiocarcinoma | interventions — lenvatinib; pembrolizumab

STUDY DESIGN:
Intervention Model Description: Patients were confirmed with advanced hepatobiliary malignancies by imaging and histological examination and meet with the inclusive criteria, including hepatocellular carcinoma, cholangiocarcinoma, ampullary carcinoma, gallbladder carcinoma, and mixed cancer)
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Lenvatinib plus Pembrolizumab (Experimental): Lenvatinib is a novel angiogenesis inhibitor which targets vascular endothelial growth factor 1-3, fibroblast growth factor receptor 1-4, platelet-derived growth factor receptor β, RET and KIT.
  Pembrolizumab is a recombinant anti-human PD-1 monoclonal antibody.
  Interventions: Drug: Lenvatinib plus Pembrolizumab

INTERVENTIONS:
Drug: Lenvatinib plus Pembrolizumab — Lenvatinib 12mg, once a day, oral at least 38 days of each 6 weeks cycle. Pembrolizumab 200mg, every 3 weeks, intravenous infused of each 6 weeks cycle. Number of cycle: until progression or unacceptable toxicity develops.
  Other Names: Lenvatinib (Lenvima, Eisai China); Pembrolizumab (Keytruda, MSD China)

SUMMARY:
The investigators design a phase IIB clinical study to explore the efficacy and safety of lenvatinib plus pembrolizumab as a second-line treatment in patients with advanced hepatobiliary malignant tumors and to analyze potential biomarkers of therapeutic response.

DETAILED DESCRIPTION:
This trial is a single-arm, non-randomized and single-center clinical study of targeted therapy combined immunotherapy in patients with hepatobiliary malignant tumors.

It is estimated that 50 patients who met the study criteria will be enrolled in PUMCH and treated with lenvatinib and pembrolizumab. The investigators will follow up and collect subjects' data each month to evaluate the efficacy and safety of treatment, including overall survival and time to progression. Multi-omics data analysis will be used to find potential biomarkers of treatment response.

ELIGIBILITY:
Inclusion Criteria: Subjects must meet all of the following criteria

* Subjects volunteer to participate in the study and agree to sign the informed consent with good compliance and follow-up.
* Subjects are 18 years old or older when signing the informed consent and gender is not limited.
* Subjects were diagnosed with advanced hepatobiliary malignant tumors (clinical stage IV) by imaging and histological examination, including hepatocellular carcinoma, cholangiocarcinoma, ampullary carcinoma, gallbladder carcinoma and mixed carcinoma.
* The disease is not suitable for radical surgery and/or topical treatment, or disease progression occurs after surgery and/or local treatment.
* At least one measurable lesion (according to RECIST version 1.1): the measurable lesion has a long diameter ≥ 10 mm or lymphadenpathy has a short diameter ≥ 15 mm in spiral CT scan.
* Patients fail after at least one systemic failure, including surgery, intervention, radiotherapy, chemotherapy and targeted therapy and require palliative treatment.
* Definition of treatment failure: Disease progression during treatment or relapse after treatment, such as after at least once radical or palliative resection surgery, revenue recurrence or progression after intervention therapy or radiotherapy. Intervention therapy or oxaliplatin treatment must be more than 1 cycle, and molecular targeted therapy must more than ≥14 days.
* Definition of intolerance: Grade ≥IV hematologic toxicity, or grade ≥III non- hematologic toxicity, or grade ≥ II damage of heart, liver and kidney during treatment.
* The ECOG score is 0-2 within 1 week before enrollment.
* Liver function assessment: Child-Pugh Grade A or mild Grade B (≤ 7 points), BCLC stage B-C.
* More than 2 weeks from first-line system treatment failure to sign informed consent for this study, and adverse events returned to normal (NCI-CTCAE ≤ I).
* Estimated survival time ≥ 6 months.
* HBV DNA <2000 IU/ml (104 copies/ml).
* Hematology and organ function are sufficient based on the following laboratory results within 14 days prior to the treatment of this study:
* Whole blood cell examination (no blood transfusion within 14 days, no G-CSF use and no drugs use): Hb≥90g/L, ANC≥1.5×10*9/L, PLT≥80×10*9/L.
* Biochemical examination (no ALB infused within 14 days): ALB≥29 g/L, ALT and AST<5×ULN, TBIL≤1.5×ULN, creatinine≤1.5×ULN (only one of albumin and bilirubin has 2 points with Child-Pugh score).
* Tumor tissue must be available for biomarker analysis prior to the first dose of treatment, If not available, participants can consult the investigator for enrollment agreement.
* Note: If an unstained section is submitted, the new section should be submitted to the laboratory within 14 days.

Exclusion Criteria: Subjects with one or more than one of the following criteria should be excluded

* Clinical stage I-III, and/or with any of the following:
* Suitable for radical surgery,
* Or, without an assessment lesion after radical surgery,
* Or, never receive any first line treatment,
* Or, liver transplantation history or ready for liver transplantation.
* ECOG score ≥ 3 points.
* Received any topical treatment within 4 weeks prior to the study, including but not limited to surgery, radiotherapy, hepatic artery embolization, TACE, hepatic artery perfusion, radiofrequency ablation, cryoablation or percutaneous ethanol injection.
* Ascites with clinical symptoms which requires abdominal puncture or drainage therapy, or Child-Pugh score >2.
* With serious systemic diseases such as heart disease and cerebrovascular disease, and the condition is unstable or uncontrollable.
* Already known active central nervous system metastasis and/or cancerous meningitis. Subjects with stable brain metastases after previous treatment may participate as long as no radiologic evidence of progression lasts for at least four weeks prior to this trial and any neurological symptoms have returned to baseline, and no new or enlarged metastatic evidence in brain and no steroids use for at least 7 days prior to trial treatment. Cancer meningitis should be excluded regardless of clinical stability.
* Surgery was performed within 4 weeks prior to the trial and patients must be
* evaluated after wound healing.
* Hepatic and renal dysfunction evidence: jaundice, ascites, and/or bilirubin ≥ 1.5 × ULN, and/or alkaline phosphatase ≥ 3 × ULN, and/or ≥ 3 grade (CTC-AE 5.0) proteinuria (> 3.5g /24 hours), or renal failure requiring blood dialysis or peritoneal dialysis.
* Urine examination shows urinary protein ≥ ++ or 24 hours urine protein >1.0g. Persistent >2 grade (CTC-AE5.0) infection.
* History of allogeneic tissue transplantation or solid organ transplantation.
* History of active tuberculosis, such as mycobacterium tuberculosis.
* Intolerant of any drug (or any excipient) in this trial.
* Female patients who are pregnant, breastfeeding or refuse contraception.
* Known or untreated brain metastases, or patients with epilepsy who need medication treatment.
* Patients with bone metastases received palliative radiotherapy (radiation area > 5% bone marrow area) within 4 weeks prior to this study, or there were wounds, ulcers or fractures that could not be healed, or patients have organ transplantation history.
* Gastrointestinal bleeding history in the past 6 months or tendency to gastrointestinal bleeding, such as esophageal varices, local active ulceration lesions, fecal occult blood ≥ (++) (gastroscopy is required when fecal occult blood is (+)).
* Evidence or history of ≥3 grade (CTC-AE5.0) bleeding events.
* History of human immunodeficiency virus infection.
* History of hepatitis B virus or hepatitis C virus infection, and not receive regular treatment.
* Severe non-healing wounds, ulcers or fractures.
* Prior treatment with either lenvatinib or any kind of anti-PD-1, anti-PD-L1 or anti-PD-L2 drugs.
* There were no active autoimmune diseases that require systemic treatment such as disease modifying drugs, corticosteroids or immunosuppressants in the past 2 years. Alternative therapies with thyroxine, insulin or corticosteroid are not considered as systemic therapy.
* Diagnosis of immunodeficiency or systemic steroid therapy or any form of immunosuppressants therapy within 7 days prior to this study. A physiological dose of corticosteroids (no more than 7.5 mg/d prednisone or equivalent) can be approved after clinical evaluation.
* There exists drug abuse, or any medical, psychological or social condition which might affect the study, the compliance or even the safety of patients.
* Variable factors which significantly affect drug use and absorption, such as inability to swallow, chronic diarrhea and intestinal obstruction.
* Any >1 grade (CTC-AE5.0) unresolved toxicity due to previous treatment or operation, except for hair loss, anemia, and hypothyroidism.
* Vaccination of any live virus vaccine within 30 days prior to this study, except for seasonal flu vaccines without live virus.
* Previous and current evidence of pulmonary fibrosis, interstitial pneumonia, pneumoconiosis, radiation pneumonitis, drug-associated pneumonia and severe impairment of lung function.
* Received a potent CYP3A4 inhibitor treatment within 7 days prior to the study, or received a potent CYP3A4 inducer within 12 days prior to the study.
* Women with fertility agree to abstinence during the treatment period and at least 6 months after the last dose (avoiding heterosexual intercourse) or using a contraceptive method with an annual contraceptive failure rate <1%.
* If a female patient has menstruation and not reached the postmenopausal state (continuously no menstruation ≥ 12 months and no other causes), and has not undergone sterilization by removing the ovaries and/or uterus), then the patient has fertility.
* Contraceptive methods with a contraceptive failure rate <1% include bilateral tubal ligation, male sterilization, hormonal contraceptives that inhibit ovulation, hormone-releasing intrauterine devices and copper intrauterine devices.
* The reliability of sexual desire should be evaluated relative to the duration of the clinical trial and lifestyle of patient. Periodic abstinence (eg. calendar days, ovulation, symptomatic body temperature or post-ovulation methods) and in vitro ejaculation are unacceptable methods of contraception.
* Male patients agree to abstinence (no heterosexual intercourse) or use of contraceptive measures and no sperm donation, as defined below:
* When a female partner has fertility, male patients must abstinence from sex during treatment and at least 6 months after the last dose of treatment, or use condoms and other contraceptive methods with contraceptive failure rate <1%. At the same time, male patients must also agree not to donate sperm.
* When a female partner is pregnant, the male patient must abstinence or using a condom during the treatment period and at least 6 months after the last dose of treatment to prevent the fetus from being affected by the study.
* The reliability of sexual desire should be evaluated relative to the duration of the clinical trial and lifestyle of patient. Periodic abstinence (eg. calendar days, ovulation, symptomatic body temperature or post-ovulation methods) and in vitro ejaculation are unacceptable methods of contraception.
* Patients are unsuitable for participation in this research after comprehensive assessment by the researchers.
* Patients participate in another clinical study at the same time.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2019-04-20 (Actual); Primary Completion 2021-04-01 (Actual); Study Completion 2021-08-01 (Actual)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | one year
  Proportion of patients whose tumor volume has reached a predetermined value and can maintain a minimum time limit, including complete response and partial response patients.
Disease Control Rate (DCR) | one year
  Proportion of patients whose tumor volume control (reduced or enlarged) reaches a predetermined value and can maintain a minimum time limit.
Progression-free Survival (PFS) | six months
  A duration from the date of initial treatment with lenvatinib plus pembrolizumab to disease progression (defined by RECIST 1.1) or death of any cause.

SECONDARY OUTCOMES:
Overall Survival (OS) | two years
  Duration from the date of initial treatment with lenvatinib plus pembrolizumab to the date of death due to any cause.
Duration of Response (DOR) | one year
  Duration from the first time reported partial response or complete response to the first time of disease progression or death.
Stable Disease | one year
  Proportion of patients with stable disease status more than 4 months.

OTHER OUTCOMES:
Incidence of Treatment-Emergent Adverse Event | two year
  Any adverse events related with treatment with lenvatinib plus pembrolizumab.

CONTACTS AND LOCATIONS:
Overall Officials: Haitao Zhao, Prof, Study Chair — Peking Union Medical College Hospital (PUMCH)
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Global Burden of Disease Cancer Collaboration; Fitzmaurice C, Akinyemiju TF, Al Lami FH, Alam T, Alizadeh-Navaei R, Allen C, Alsharif U, Alvis-Guzman N, Amini E, Anderson BO, Aremu O, Artaman A, Asgedom SW, Assadi R, Atey TM, Avila-Burgos L, Awasthi A, Ba Saleem HO, Barac A, Bennett JR, Bensenor IM, Bhakta N, Brenner H, Cahuana-Hurtado L, Castaneda-Orjuela CA, Catala-Lopez F, Choi JJ, Christopher DJ, Chung SC, Curado MP, Dandona L, Dandona R, das Neves J, Dey S, Dharmaratne SD, Doku DT, Driscoll TR, Dubey M, Ebrahimi H, Edessa D, El-Khatib Z, Endries AY, Fischer F, Force LM, Foreman KJ, Gebrehiwot SW, Gopalani SV, Grosso G, Gupta R, Gyawali B, Hamadeh RR, Hamidi S, Harvey J, Hassen HY, Hay RJ, Hay SI, Heibati B, Hiluf MK, Horita N, Hosgood HD, Ilesanmi OS, Innos K, Islami F, Jakovljevic MB, Johnson SC, Jonas JB, Kasaeian A, Kassa TD, Khader YS, Khan EA, Khan G, Khang YH, Khosravi MH, Khubchandani J, Kopec JA, Kumar GA, Kutz M, Lad DP, Lafranconi A, Lan Q, Legesse Y, Leigh J, Linn S, Lunevicius R, Majeed A, Malekzadeh R, Malta DC, Mantovani LG, McMahon BJ, Meier T, Melaku YA, Melku M, Memiah P, Mendoza W, Meretoja TJ, Mezgebe HB, Miller TR, Mohammed S, Mokdad AH, Moosazadeh M, Moraga P, Mousavi SM, Nangia V, Nguyen CT, Nong VM, Ogbo FA, Olagunju AT, Pa M, Park EK, Patel T, Pereira DM, Pishgar F, Postma MJ, Pourmalek F, Qorbani M, Rafay A, Rawaf S, Rawaf DL, Roshandel G, Safiri S, Salimzadeh H, Sanabria JR, Santric Milicevic MM, Sartorius B, Satpathy M, Sepanlou SG, Shackelford KA, Shaikh MA, Sharif-Alhoseini M, She J, Shin MJ, Shiue I, Shrime MG, Sinke AH, Sisay M, Sligar A, Sufiyan MB, Sykes BL, Tabares-Seisdedos R, Tessema GA, Topor-Madry R, Tran TT, Tran BX, Ukwaja KN, Vlassov VV, Vollset SE, Weiderpass E, Williams HC, Yimer NB, Yonemoto N, Younis MZ, Murray CJL, Naghavi M. Global, Regional, and National Cancer Incidence, Mortality, Years of Life Lost, Years Lived With Disability, and Disability-Adjusted Life-Years for 29 Cancer Groups, 1990 to 2016: A Systematic Analysis for the Global Burden of Disease Study. JAMA Oncol. 2018 Nov 1;4(11):1553-1568. doi: 10.1001/jamaoncol.2018.2706. PMID 29860482
- [Background] Kamangar F, Dores GM, Anderson WF. Patterns of cancer incidence, mortality, and prevalence across five continents: defining priorities to reduce cancer disparities in different geographic regions of the world. J Clin Oncol. 2006 May 10;24(14):2137-50. doi: 10.1200/JCO.2005.05.2308. PMID 16682732
- [Background] Ferlay J, Soerjomataram I, Dikshit R, Eser S, Mathers C, Rebelo M, Parkin DM, Forman D, Bray F. Cancer incidence and mortality worldwide: sources, methods and major patterns in GLOBOCAN 2012. Int J Cancer. 2015 Mar 1;136(5):E359-86. doi: 10.1002/ijc.29210. Epub 2014 Oct 9. PMID 25220842
- [Background] Ryerson AB, Eheman CR, Altekruse SF, Ward JW, Jemal A, Sherman RL, Henley SJ, Holtzman D, Lake A, Noone AM, Anderson RN, Ma J, Ly KN, Cronin KA, Penberthy L, Kohler BA. Annual Report to the Nation on the Status of Cancer, 1975-2012, featuring the increasing incidence of liver cancer. Cancer. 2016 May 1;122(9):1312-37. doi: 10.1002/cncr.29936. Epub 2016 Mar 9. PMID 26959385
- [Background] Yamamoto Y, Matsui J, Matsushima T, Obaishi H, Miyazaki K, Nakamura K, Tohyama O, Semba T, Yamaguchi A, Hoshi SS, Mimura F, Haneda T, Fukuda Y, Kamata JI, Takahashi K, Matsukura M, Wakabayashi T, Asada M, Nomoto KI, Watanabe T, Dezso Z, Yoshimatsu K, Funahashi Y, Tsuruoka A. Lenvatinib, an angiogenesis inhibitor targeting VEGFR/FGFR, shows broad antitumor activity in human tumor xenograft models associated with microvessel density and pericyte coverage. Vasc Cell. 2014 Sep 6;6:18. doi: 10.1186/2045-824X-6-18. eCollection 2014. PMID 25197551
- [Background] Kudo M, Finn RS, Qin S, Han KH, Ikeda K, Piscaglia F, Baron A, Park JW, Han G, Jassem J, Blanc JF, Vogel A, Komov D, Evans TRJ, Lopez C, Dutcus C, Guo M, Saito K, Kraljevic S, Tamai T, Ren M, Cheng AL. Lenvatinib versus sorafenib in first-line treatment of patients with unresectable hepatocellular carcinoma: a randomised phase 3 non-inferiority trial. Lancet. 2018 Mar 24;391(10126):1163-1173. doi: 10.1016/S0140-6736(18)30207-1. PMID 29433850
- [Background] Sprinzl MF, Galle PR. Current progress in immunotherapy of hepatocellular carcinoma. J Hepatol. 2017 Mar;66(3):482-484. doi: 10.1016/j.jhep.2016.12.009. Epub 2016 Dec 21. No abstract available. PMID 28011330
- [Background] Topalian SL, Drake CG, Pardoll DM. Immune checkpoint blockade: a common denominator approach to cancer therapy. Cancer Cell. 2015 Apr 13;27(4):450-61. doi: 10.1016/j.ccell.2015.03.001. Epub 2015 Apr 6. PMID 25858804
- [Background] Rotte A, Jin JY, Lemaire V. Mechanistic overview of immune checkpoints to support the rational design of their combinations in cancer immunotherapy. Ann Oncol. 2018 Jan 1;29(1):71-83. doi: 10.1093/annonc/mdx686. PMID 29069302
- [Background] Jia Y, Zeng Z, Li Y, Li Z, Jin L, Zhang Z, Wang L, Wang FS. Impaired function of CD4+ T follicular helper (Tfh) cells associated with hepatocellular carcinoma progression. PLoS One. 2015 Feb 17;10(2):e0117458. doi: 10.1371/journal.pone.0117458. eCollection 2015. PMID 25689070
- [Background] Zhu AX, Finn RS, Edeline J, Cattan S, Ogasawara S, Palmer D, Verslype C, Zagonel V, Fartoux L, Vogel A, Sarker D, Verset G, Chan SL, Knox J, Daniele B, Webber AL, Ebbinghaus SW, Ma J, Siegel AB, Cheng AL, Kudo M; KEYNOTE-224 investigators. Pembrolizumab in patients with advanced hepatocellular carcinoma previously treated with sorafenib (KEYNOTE-224): a non-randomised, open-label phase 2 trial. Lancet Oncol. 2018 Jul;19(7):940-952. doi: 10.1016/S1470-2045(18)30351-6. Epub 2018 Jun 3. PMID 29875066
- [Background] Le DT, Uram JN, Wang H, Bartlett BR, Kemberling H, Eyring AD, Skora AD, Luber BS, Azad NS, Laheru D, Biedrzycki B, Donehower RC, Zaheer A, Fisher GA, Crocenzi TS, Lee JJ, Duffy SM, Goldberg RM, de la Chapelle A, Koshiji M, Bhaijee F, Huebner T, Hruban RH, Wood LD, Cuka N, Pardoll DM, Papadopoulos N, Kinzler KW, Zhou S, Cornish TC, Taube JM, Anders RA, Eshleman JR, Vogelstein B, Diaz LA Jr. PD-1 Blockade in Tumors with Mismatch-Repair Deficiency. N Engl J Med. 2015 Jun 25;372(26):2509-20. doi: 10.1056/NEJMoa1500596. Epub 2015 May 30. PMID 26028255
- [Background] Le DT, Durham JN, Smith KN, Wang H, Bartlett BR, Aulakh LK, Lu S, Kemberling H, Wilt C, Luber BS, Wong F, Azad NS, Rucki AA, Laheru D, Donehower R, Zaheer A, Fisher GA, Crocenzi TS, Lee JJ, Greten TF, Duffy AG, Ciombor KK, Eyring AD, Lam BH, Joe A, Kang SP, Holdhoff M, Danilova L, Cope L, Meyer C, Zhou S, Goldberg RM, Armstrong DK, Bever KM, Fader AN, Taube J, Housseau F, Spetzler D, Xiao N, Pardoll DM, Papadopoulos N, Kinzler KW, Eshleman JR, Vogelstein B, Anders RA, Diaz LA Jr. Mismatch repair deficiency predicts response of solid tumors to PD-1 blockade. Science. 2017 Jul 28;357(6349):409-413. doi: 10.1126/science.aan6733. Epub 2017 Jun 8. PMID 28596308
- [Background] Ma WJ, Wang HY, Teng LS. Correlation analysis of preoperative serum alpha-fetoprotein (AFP) level and prognosis of hepatocellular carcinoma (HCC) after hepatectomy. World J Surg Oncol. 2013 Aug 27;11:212. doi: 10.1186/1477-7819-11-212. PMID 23981851
- [Background] Asano M. Hepatectomy and arterial blood ketone-body ratio. II. Clinical significance of arterial blood ketone-body ratio in hepatectomized patients. Nihon Geka Hokan. 1984 May 1;53(3):485-96. No abstract available. PMID 6095784
- [Background] Gao Q, Wang XY, Qiu SJ, Yamato I, Sho M, Nakajima Y, Zhou J, Li BZ, Shi YH, Xiao YS, Xu Y, Fan J. Overexpression of PD-L1 significantly associates with tumor aggressiveness and postoperative recurrence in human hepatocellular carcinoma. Clin Cancer Res. 2009 Feb 1;15(3):971-9. doi: 10.1158/1078-0432.CCR-08-1608. PMID 19188168
- [Background] El-Khoueiry AB, Sangro B, Yau T, Crocenzi TS, Kudo M, Hsu C, Kim TY, Choo SP, Trojan J, Welling TH Rd, Meyer T, Kang YK, Yeo W, Chopra A, Anderson J, Dela Cruz C, Lang L, Neely J, Tang H, Dastani HB, Melero I. Nivolumab in patients with advanced hepatocellular carcinoma (CheckMate 040): an open-label, non-comparative, phase 1/2 dose escalation and expansion trial. Lancet. 2017 Jun 24;389(10088):2492-2502. doi: 10.1016/S0140-6736(17)31046-2. Epub 2017 Apr 20. PMID 28434648
- [Background] Soyano AE, Dholaria B, Marin-Acevedo JA, Diehl N, Hodge D, Luo Y, Manochakian R, Chumsri S, Adjei A, Knutson KL, Lou Y. Peripheral blood biomarkers correlate with outcomes in advanced non-small cell lung Cancer patients treated with anti-PD-1 antibodies. J Immunother Cancer. 2018 Nov 23;6(1):129. doi: 10.1186/s40425-018-0447-2. PMID 30470260
- [Background] Snyder A, Makarov V, Merghoub T, Yuan J, Zaretsky JM, Desrichard A, Walsh LA, Postow MA, Wong P, Ho TS, Hollmann TJ, Bruggeman C, Kannan K, Li Y, Elipenahli C, Liu C, Harbison CT, Wang L, Ribas A, Wolchok JD, Chan TA. Genetic basis for clinical response to CTLA-4 blockade in melanoma. N Engl J Med. 2014 Dec 4;371(23):2189-2199. doi: 10.1056/NEJMoa1406498. Epub 2014 Nov 19. PMID 25409260
- [Background] Gately MK, Warrier RR, Honasoge S, Carvajal DM, Faherty DA, Connaughton SE, Anderson TD, Sarmiento U, Hubbard BR, Murphy M. Administration of recombinant IL-12 to normal mice enhances cytolytic lymphocyte activity and induces production of IFN-gamma in vivo. Int Immunol. 1994 Jan;6(1):157-67. doi: 10.1093/intimm/6.1.157. PMID 7908534
- [Background] Frucht DM, Fukao T, Bogdan C, Schindler H, O'Shea JJ, Koyasu S. IFN-gamma production by antigen-presenting cells: mechanisms emerge. Trends Immunol. 2001 Oct;22(10):556-60. doi: 10.1016/s1471-4906(01)02005-1. PMID 11574279
- [Background] Shin T, Nakayama T, Akutsu Y, Motohashi S, Shibata Y, Harada M, Kamada N, Shimizu C, Shimizu E, Saito T, Ochiai T, Taniguchi M. Inhibition of tumor metastasis by adoptive transfer of IL-12-activated Valpha14 NKT cells. Int J Cancer. 2001 Feb 15;91(4):523-8. doi: 10.1002/1097-0215(20010215)91:43.0.co;2-l. PMID 11251976
- [Background] Schroder K, Hertzog PJ, Ravasi T, Hume DA. Interferon-gamma: an overview of signals, mechanisms and functions. J Leukoc Biol. 2004 Feb;75(2):163-89. doi: 10.1189/jlb.0603252. Epub 2003 Oct 2. PMID 14525967
- [Background] Lee IC, Huang YH, Chau GY, Huo TI, Su CW, Wu JC, Lin HC. Serum interferon gamma level predicts recurrence in hepatocellular carcinoma patients after curative treatments. Int J Cancer. 2013 Dec 15;133(12):2895-902. doi: 10.1002/ijc.28311. Epub 2013 Jun 25. PMID 23749461
- [Result] Lin J, Yang X, Long J, Zhao S, Mao J, Wang D, Bai Y, Bian J, Zhang L, Yang X, Wang A, Xie F, Shi W, Yang H, Pan J, Hu K, Guan M, Zhao L, Huo L, Mao Y, Sang X, Wang K, Zhao H. Pembrolizumab combined with lenvatinib as non-first-line therapy in patients with refractory biliary tract carcinoma. Hepatobiliary Surg Nutr. 2020 Aug;9(4):414-424. doi: 10.21037/hbsn-20-338. PMID 32832493